CLINICAL TRIAL: NCT01794663
Title: A Three-Part, Multi-Centre, Randomised, Double-Blind, Placebo-Controlled, Parallel-Group, Sequential Adaptive, Phase II Study to Evaluate the Safety, Tolerability and Efficacy of OPN-305, a Humanised Monoclonal Antibody That Blocks Toll-Like Receptor 2, in Renal Transplant Patients at High Risk of Delayed Graft Function
Brief Title: Placebo-Controlled Study to Evaluate the Safety and Efficacy of OPN-305 in Preventing Delayed Renal Graft Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Opsona Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OPN305-102; 2012-001455-39 (EudraCT Number)
Record Dates: First submitted 2013-02-13; First posted 2013-02-20 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2017-02

CONDITIONS: Delayed Graft Function
Keywords: Early kidney graft dysfunction; renal transplantation
MeSH Terms: conditions — Delayed Graft Function | interventions — tomaralimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OPN-305 (Experimental)
  Interventions: Drug: OPN-305
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OPN-305 — Intravenous infusion for 1 hour at start of transplant procedure
  Arms: OPN-305
Drug: Placebo — Intravenous infusion for 1 hour at start of transplant procedure
  Arms: Matching placebo

SUMMARY:
When a patient receives a kidney transplant particularly if the kidney is from an older donor or one who has had the kidney removed after their heart has stopped, there is a risk that the newly transplanted kidney may not function immediately. If the delay in function means that dialysis is needed in the first 7 days after the transplantation then this is known as delayed graft function or dDGF. Also delayed graft function that does not require dialysis but is present because the serum creatinine does not fall sufficiently is known as functional delayed graft function or fDGF. This problem is often due to an excessive inflammatory reaction to not having had a blood supply between the time of donation and transplant.

OPN-305 is a monoclonal antibody that blocks Toll-like Receptor 2 which is thought to be partly responsible for increasing the risk of this inflammation. It is hoped that the effects of the inflammation will be reduced and therefore prevent dDGF and fDGF from occurring.

The purpose of the study is to explore how effective OPN-305 is in preventing dDGF and fDGF as well as improving other measures of kidney function and the overall safety of the antibody. In the first part of the study, each patient received an Infusion of one of three possible doses of OPN-305 or a placebo and in the second part the most suitable dose of OPN-305 and a placebo would be used. The purpose of this second part of the study is to find out if a dose of OPN-305 which has already been tested in an earlier part of this study can prevent kidney graft dysfunction. For the purposes of this study, kidney function will be assessed using the composite of delayed graft function (dDGF) because dialysis is necessary in the first 7 days and functional delayed graft function that does not require dialysis but is present because the serum creatinine, a key measure of renal function, does not fall sufficiently (fDGF) in the first 7 days post-transplant.

Protocol OPN305-103 follows out to 12 months post-transplant the clinical status and graft function of patients who have completed the 6-month post-transplant period under Part A or Part B of OPN305-102.

ELIGIBILITY:
Inclusion criteria

INCLUSION CRITERIA FOR TRANSPLANT RECIPIENTS

* First or second renal transplant recipient - for second renal transplantations;

  * The second transplant should NOT be due to rejection
  * Panel Reactive Antibody (PRA) should be <10%
  * Minimum 3 months since the loss of the first transplanted kidney
* Dialysis-dependent at the time of transplantation as documented by:

  * Requirement for at least 2 dialysis sessions/week in the 56 days before transplantation

INCLUSION CRITERIA FOR DONOR KIDNEY:

* The donor kidney must be considered compatible according to local transplant guidelines
* An ECD donor defined as:

  o Extended Criteria Donor defined as:
  * Donor ≥60 years of age
  * Donor 50-59 years of age with two of three of the following criteria present:
  * Death due to cerebrovascular accident
  * Pre-existing history of systemic hypertension
  * Terminal creatinine > 1.5mg/dL (132.6 µmol/L)
* Kidney allograft maintained in cold storage with or without machine perfusion

Exclusion Criteria

EXCLUSION CRITERIA FOR TRANSPLANT RECIPIENTS:

* Use of an investigational drug in the 30 days before Study Day 1
* Participation in any other research
* Known hypersensitivity to human monoclonal antibodies or any of the study-drug excipients
* Previous hypersensitivity to basiliximab or anti-thymocyte globulin (ATG)
* History or known HIV, HBV, or HCV-positive
* History of malignancy within the last five years, except excised squamous or basal cell carcinoma of the skin or cervical intraepithelial neoplasia
* Scheduled to undergo multi-organ transplantation
* Planned dual kidney transplantation
* Presence of clinically significant infections requiring continued therapy
* Active tuberculosis
* Existence of any surgical or medical condition, other than the current transplantation which, in the opinion of the investigator, might significantly alter the distribution, metabolism or excretion of study medication
* Presence of uncontrolled diabetes mellitus.
* Current drug and/or alcohol abuse
* History or presence of a medical condition or disease that in the investigator's assessment would place the patient at an unacceptable risk for study participation
* Lactating or pregnant woman
* Patient institutionalized by administrative or court order

EXCLUSION CRITERIA FOR ALL DONOR KIDNEYS

* DCD or SCD donor kidney
* Terminal creatinine >3mg/dL
* Donor who is known to have received an investigational drug for I-R injury or graft rejection (immunosuppressant) in the 48h before organ recovery
* Participation in any other research (drug or non-drug)
* Kidney donor <5 years of age or <20kg body weight
* Living donor allograft
* HLA or ABO incompatible kidney as defined by a negative cytotoxic crossmatch
* Donor institutionalized by administrative or court order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2012-10; Primary Completion 2016-06-30 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Measure of Early Graft Function EGF | First 7 days following renal transplantation
  Initiation of dialysis in the first 7 days following renal transplantation and failure of serum creatinine to decrease by at least 10% daily on 3 successive days during the first week post transplantation

SECONDARY OUTCOMES:
Creatinine at 7 and 14 days and at 1, 3 and 6 months | 7 and 14 days and at 1, 3 and 6 months
  Measure of creatinine at 7 and 14 days and at 1, 3 and 6 months
Cystatin C at 7 and 14 days and at 1, 3 and 6 months | 7 and 14 days and at 1, 3 and 6 months
  Measure of Cystatin C at 7 and 14 days and at 1, 3 and 6 months
Symmetrical dimethylarginine at 7 and 14 days and at 1, 3 and 6 months | 7 and 14 days and at 1, 3 and 6 months
  Measure of symmetrical dimethylarginine at 7 and 14 days and at 1, 3 and 6 months
Incidence of slow graft function | 5 days post-transplant
  Slow graft function to be assessed over first 5 days post-transplant
Serum creatinine over time | over the duration of follow-up
  Measure of Serum creatinine over time
Composite endpoint | 6 months
  Components of the composite endpoint are:
  1. Incidence of biopsy-proven kidney allograft rejection (biopsies will be done on a for-cause basis only)
  2. Graft loss
  3. Reports of patient death(s)
  4. Patients lost to follow-up
Time to biopsy-proven kidney allograft rejection | 6 months
  Time to biopsy-proven kidney allograft rejection
Time to first dialysis or functional delayed graft function and delayed graft function duration | 30 days
  Duration of DGF is defined as either:
  Time from transplantation to time of completion of final dialysis for DGF
  Time from transplantation to time when creatinine starts to fall by at least 10% without dialysis
Blood and urine biomarkers for acute kidney injury (AKI) | days 2, 7, 14, 28, 90 and 180
  Serum NGAL, urinary NGAL, α-GST, π-GST, KIM-1 and IL-18
Duration of initial hospitalization | 6 months
  Duration of initial hospitalization
Duration of subsequent readmissions | 6 months
  Duration of subsequent readmissions
Reason for subsequent readmissions | 6 months
  Reason for subsequent readmissions
Number of Adverse events (AEs) | 6 months
  Number of Adverse events (AEs)
Nature of Adverse events (AEs) | 6 months
  Nature of Adverse events (AEs)
Incidence of infections | 6 months
  Incidence of infections by category and organism
Rate of primary non-function (permanent lack of function of the allograft) | 6 months
Number of dialysis sessions between 0 and 30 days post-transplantation | 30 days
  Number of dialysis sessions between 0 and 30 days post-transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Miller, FRCS MBBS, Study Director — OpsonaTherapeutics Ltd.
Locations (45):
- United States (13):
  - Research Site, Los Angeles, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Site, New Orleans, Louisiana
  - Research Site, Livingston, New Jersey
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Harrisburg, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Richmond, Virginia
- Research Site, Linz, Austria
- Belgium (4):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Liège
- Research Site, Prague, Czechia
- France (3):
  - Research Site, Bordeaux
  - Research Site, Paris
  - Research Site, Toulouse
- Germany (9):
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Erlangen
  - Research Site, Heidelberg
  - Research Site, Mannheim
  - Research Site, Münster
  - Research Site, Tübingen
- Netherlands (4):
  - Research Site, Groningen
  - Research Site, Leiden
  - Research Site, Nijmegen
  - Research Site, Rotterdam
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Lodz
  - Research Site, Szczecin
  - Research Site, Warsaw
- Spain (3):
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Santander
- Research Site, Zurich, Switzerland
- United Kingdom (2):
  - Research Site, London
  - Research Site, Newcastle upon Tyne